CLINICAL TRIAL: NCT02362906
Title: Assessing the Effectiveness of Integrative Treatment That Combines Interior and Exterior Treatment Plans in Pediatric Pneumonia: a Program by the Special Scientific Research Fund of Public Welfare Profession of China
Brief Title: Effectiveness Study of Integrative Treatment for Pediatric Community Acquired Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liaoning University of Traditional Chinese Medicine (Other)
Collaborators: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xuefeng Wang, Chief physician, Liaoning University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201307007
Record Dates: First submitted 2015-01-22; First posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Pneumonia
Keywords: pneumonia; pediatrics
MeSH Terms: conditions — Pneumonia | interventions — Second Generation Cephalosporins; Erythromycin; Azithromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Injection,medications and application (Experimental): Intravenous injection:
  bacterial pneumonia: second generation cephalosporin; mycoplasma pneumonia: erythromycin or azithromycin; viral pneumonia: Xiyanping injection, produced by Jiangxi Qing Feng Pharmaceutical Co.,Ltd; Medications: according to TCM syndrome differentiations; Wind-heat blocking lungs pattern(feng re bi fei zheng): wind-heat formula granules; phlegm-heat blocking lungs pattern(tan re bi fei zheng): phlegm-heat formula granules; external application: Fu-xiong San.
  Interventions: Drug: Xiyanping injection; Drug: wind-heat formula granules; Drug: phlegm-heat formula granules; Drug: Fu-xiong San; Drug: second generation cephalosporin; Drug: Erythromycin; Drug: Azithromycin
- Injection and medications (Experimental): Intravenous injection:
  bacterial pneumonia：second generation cephalosporin; mycoplasma pneumonia：erythromycin or azithromycin; viral pneumonia：Xiyanping injection, produced by Jiangxi Qing Feng Pharmaceutical Co.,Ltd; Medications: according to TCM syndrome differentiations; Wind-heat blocking lungs pattern(feng re bi fei zheng): wind-heat formula granules; phlegm-heat blocking lungs pattern(tan re bi fei zheng): phlegm-heat formula granules.
  Interventions: Drug: Xiyanping injection; Drug: wind-heat formula granules; Drug: phlegm-heat formula granules; Drug: second generation cephalosporin; Drug: Erythromycin; Drug: Azithromycin
- Injection and application (Experimental): Intravenous injection:
  bacterial pneumonia: second generation cephalosporin; mycoplasma pneumonia: erythromycin or azithromycin; viral pneumonia: Xiyanping injection, produced by Jiangxi Qing Feng Pharmaceutical Co.,Ltd; external application: Fu-xiong San.
  Interventions: Drug: Xiyanping injection; Drug: Fu-xiong San; Drug: second generation cephalosporin; Drug: Erythromycin; Drug: Azithromycin

INTERVENTIONS:
Drug: Xiyanping injection — ivd. 5 to 10 mg/(kg•d), plus 5% Glucose Injection, 80 to 100 ml, ivd. Once a day injection
Drug: wind-heat formula granules — children aged 6 months to 3-year old: 1/2 packet，orally taken two times daily or frequency; children aged 3 to 5-year old: 2/3 packet，orally taken two times daily or frequency; children aged 5 to 14-year old: 1 packet， orally taken two times daily or frequency
  Arms: Injection and medications; Injection,medications and application
Drug: phlegm-heat formula granules — children aged 6 months to 3-year old: 1/2 packet，orally taken two times daily or frequency; children aged 3 to 5-year old: 2/3 packet，orally taken two times daily or frequency; children aged 5 to 14-year old: 1 packet， orally taken two times daily or frequency
  Arms: Injection and medications; Injection,medications and application
Drug: Fu-xiong San — external application; 8-10 cm wide, 0.3-0.5 cm thick;10 mins for patient aged 1 to 3-year old; 15 mins for those aged 3 to 5-year old; once daily
  Arms: Injection and application; Injection,medications and application
Drug: second generation cephalosporin
Drug: Erythromycin — ivd. 30 mg/(kg•d), plus 5% Glucose Injection, 80 to 500 ml, ivd. Once a day injection
Drug: Azithromycin — ivd. 10 mg/(kg•d), plus 5% Glucose Injection, 100 to 500 ml, ivd. Once a day injection

SUMMARY:
The purpose of this study is to evaluate the effectiveness of traditional Chinese medicine for treatment of pediatric pneumonia. It is a multicenter randomized controlled trial.

DETAILED DESCRIPTION:
The block randomization is used in this trial. Random numbers are generated by statistical analysis system(SAS) software. Statistical analysis staff and those who perform the follow-up are blinded. Sample size calculation was performed, which was 1164 , and considering drop-out or withdrawal, investigators plan to enroll 1500 patients (500 in experimental group 1, 500 in experimental group 2, 500 in experimental group 3).

ELIGIBILITY:
Inclusion Criteria:

* children,aged 1 to 14 years old;
* diagnosed as pneumonia according to western medicine diagnostic criteria;
* diagnosed as TCM pneumonia with pneumonia with dyspnea and cough, meeting wind-heat blocking lungs pattern (feng re bi fei zheng), and phlegm-heat blocking lungs pattern(tan re bi fei zheng);
* disease progression within 72 hours; those whose guardians understood and assigned the informed consent;

Exclusion Criteria:

* severe pneumonia;
* complicated with other Pulmonary Disorders attack other than pneumonia;
* complicated with primary disease of heart(congenital heart disease, myocarditis, et al),liver(alanine aminotransferase(ALT),and aspartate transaminase(AST) ≥1.5 times of normal value ceiling),kidney (blood urea nitrogen(BUN) >8.2mmol/l, or serum C reactive protein >104umol/l,et al) and blood system (anemia) ,and those with psychopathy;
* allergic to interventional medications; those who are participating or have participated in other clinical trials in 3 months;
* those who intend to lost follow-up by practitioners' judgment.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Cured rate (clinical symptoms and signs totally disappear, the period of lab tests return to normal is recorded) | every day since receiving treatment,all together 7 days (times)
  clinical symptoms and signs totally disappear, the period of lab tests return to normal is recorded
effective time window (days range from treatment is received to the effectiveness is observed, and symptoms disappear) | every day since receiving treatment, all together 7 days (times)
  days range from treatment is received to the effectiveness is observed, and symptoms disappear

SECONDARY OUTCOMES:
effect in treating fever | 7 days
  temperature, fever frequency,fever lasting time, Ibuprofen Suspension， all to be measured
effect in dyspnea releasing | 7 days
  gasp frequency, severity, all to be measured
effect in phlegm releasing | 7 days
  phlegm amount,color and nature to be measured
effect in cough releasing | 7 days
  cough severity to be measured
time from admission to recovery of rales | 7 days
TCM syndrome scores | 7 days
  measure is a composite.
effective rate of TCM syndrome scores | 7 days
  total effecive rate according to TCM syndrome differentiation and treatment, and single syndrome effective rate
check-out time (days counted when the patient checks out) | 7 days
  days counted when the patient checks out
pulmonary disease incidence (prolonged pneumonia, chronic cough, cough variant asthma incidence in the follow-up) | 15 days; 30 days; 90 days
  prolonged pneumonia, chronic cough, cough variant asthma incidence in the follow-up
safety (With adverse events as the calculation basis) | 7 days
  With adverse events as the calculation basis

OTHER OUTCOMES:
direct medical cost | observed during treatment in 7 days
  medical cost including hospital expenses, examine fee, medication fee, et al, relate to treatment in hospital

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Affiliated Children's Hospital of Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Guangzhou Children's Hospital, Guangzhou, Guangdong
  - Affiliated hospital of Guangzhou university of Chinese Medicine, Guangzhou, Guangdong
  - Affiliated Hospital of Guangxi University of Chinese Medicine, Nanning, Guangxi
  - Affiliated Hospital of Changchun University of TCM, Changchun, Jilin
  - Affiliated Children's Hospital of Dalian Medical University, Dalian, Liaoning
  - Affiliated Hospital of Liaoning University of TCM, Shenyang, Liaoning
  - Affiliated Hospital of Shandong University of TCM, Ji'nan, Shandong
  - Affiliated Longhua Hospital of Shanghai University of TCM, Shanghai, Shanghai Municipality
  - First teaching hospital of Tianjin university of TCM, Tianjin, Tianjin Municipality